CLINICAL TRIAL: NCT04674618
Title: Ultrasound-assisted vs Landmark Based Intrathecal Administration of Nusinersen in Adult Patients With SMA Disease: a Randomized Trial
Brief Title: Ultrasound-assisted vs Landmark Based Intrathecal Administration of Nusinersen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3352
Record Dates: First submitted 2020-12-10; First posted 2020-12-19 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2021-07

CONDITIONS: Muscular Atrophy, Spinal; Ultrasound
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- US-assisted nusinersen administration (Experimental): A paramedian sagittal oblique view will be used to identify with ultrasound specific lumbar interspaces. After local anesthesia the spinal needle will be used to identify subarachnoid space. After confirmation of the flow of cerebrospinal fluid and after removing 5 ml of CSF, nusinersen will be administered intrathecally over 1-3 min.
  Interventions: Device: US-assisted nusinersen administration
- landmark based nusinersen administration (No Intervention): The desired intervertebral space will be first identified by manual palpation of surface landmarks and marked on the skin. After local anesthesia the spinal needle will be usedto identify subarachnoid space. After confirmation of the flow of cerebrospinal fluid and after removing 5 ml of CSF, nusinersen will be administered intrathecally over 1-3 min.

INTERVENTIONS:
Device: US-assisted nusinersen administration — Ultrasound identification of intervertebral space (L2-L3 or L3-L4)
  Arms: US-assisted nusinersen administration

SUMMARY:
Intrathecal administration of Nusinersen, an antisense oligonucleotide capable of increasing Survival Motor Neuron protein production, has been tested in Spinal Muscular Atrophy (SMA) to improve motor function and survival. A feature of adult SMA patients is a progressive neuromyopathic scoliosis, so spinal nusinersen administration can be challenging. Landmark identification using a pre-procedure ultrasound (US) facilitates technical performance of spinal anesthesia and allows for the elimination of radiation exposure.

The aim of this randomized prospectic study is to determine if the US assistance for spinal administration of nusinersen is able to increase the proportion at successful 1st needle insertion of the needle. Secondary outcome measures are procedure time, patient satisfaction and prevalence of postdural puncture headache.

Patients will be randomlized to receive a US-assisted nusinersen administration or a landmark based nusinersen administration.

DETAILED DESCRIPTION:
Background Nusinersen, an antisense oligonucleotide (ASO) capable of increasing SMN protein production, has been used in clinical trials in infants and children with SMA type 1 or type 2 and has been associated to a significantly better motor development, motor function, and survival compared with placebo groups. Because of the lacking ability of ASOs to cross the blood-brain barrier, nusinersen is administered intrathecally. While most infants with SMA type 1 die in easy childhood without a muscular and nutritional support, SMA type 2 patients often reach adulthood, and patients with SMA type 3 generally have a normal lifespan. A further feature of SMA patients is a progressive neuromyopathic scoliosis, so spinal nusinersen administration can be challenging because of poorly palpable surface landmarks, as in elderly and in obese patients. In patients with anticipated difficult anatomy, the failure rate of neuraxial anesthesia may be as high as 17%. Furthermore, multiple needle punctures are associated with hematoma, post-dural-puncture headache, back pain, and patient dissatisfaction. Current data suggest that landmark identification using a pre-procedure ultrasound (US) is a useful adjunct to neuraxial anesthesia that facilitates technical performance in obstetric and pediatric patients. In adult patients with difficult spinal anatomy a pre-procedure US reduces the number of attempts and the number of needle passes necessary for successful spinal anesthesia and can predict technical difficulty; notably, compared to fluoroscopy, sonography allows for the elimination of radiation exposure for patient and physician and for a cost reduction for institution. Despite these potential advantages, reports of lumbar central neuraxial blocks US guidance in patients with predicted placement difficulties are limited. Most reports to date involve a small number of patients with normal anatomy.

Methods The study will be conducted in Fondazione Policlinico "A.Gemelli" operatory rooms, Rome, Italy. Written informed consent will be obtained from all patients enrolled in the study. SMA adult patients referring to NEMO center of this institution will be enrolled. Exclusion criteria will be: coagulation defects, patients medicated with anticoagulation, any finding of infection in puncture site, high intracranial pressure. A visit will be performed before the procedure.

Patients will be randomly assigned in ratio 1:1 to one of two groups using a sealed envelope: Group 1 (US-assisted nusinersen administration) and Group 2 (landmark based nusinersen administration). Nusinersen administration will be performed with a single-operator technique by one of two anesthesiologists trained on US-guided or -assisted central neuraxial blocks. With patient in sitting position, or in lateral position if forced posture will be needed, after skin disinfection with 2% chlorhexidine in 70% alcohol, the spinal administration will be performed as follows: Group 1 (US- guided nusinersen administration). The paramedian sagittal oblique view will be used to identify specific lumbar interspaces and perform the procedure. Starting at the sacrum and moving cephalad, the L2-3 or L3-4 intervertebral interspace will be identified. After local anesthesia with lidocaine 2% (3-5 mL), a 25-gauge Withacre spinal needle will be used to identify subarachnoid space. After confirmation of the flow of cerebrospinal fluid and after removing 5 ml of CSF, nusinersen will be administered intrathecally over 1-3 min. Group 2 (landmark based nusinersen administration).

The desired intervertebral space (L2-3 or L3-4) was first identified by manual palpation of surface landmarks and marked on the skin. After local anesthesia with lidocaine 2% (3-5 mL) a 25-gauge Withacre spinal needle will be used. After confirmation of the flow of cerebrospinal fluid and after removing 5 ml of CSF, nusinersen will be administered as previously described. After successful administration, patients will be positioned in the supine position for 2-3 h. Within 72 hours of administration a phone survey will be conducted to evaluate the development of postdural puncture headache. Another outpatient visit will be performed at 30 days after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* SMA adult patients

Exclusion Criteria:

* coagulation defects;
* medication with anticoagulant;
* infection in puncture site;
* high intracranial pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Number of attempts | During the procedure (spinal injection of nusinersen)
  The number of needle insertions through the skin surface. If complete withdrawal of the needle from the patient's skin surface will be needed, followed by reinsertion in a different skin location or a different spinal level, this will be counted as a second attempt.

SECONDARY OUTCOMES:
Successful administration | During the procedure (spinal injection of nusinersen)
  confirmation of the flow of cerebrospinal fluid through the spinal needle and subsequent nusinersen administration
Procedure time | During the procedure (spinal injection of nusinersen)
  the time in seconds from the start of US imaging to visualization of cerebrospinal fluid flow in intervention group and from the first hand contact to the skin to visualization of cerebrospinal fluid flow in control group.
Patients satisfaction | 5 minutes after the end of the procedure (spinal injection of nusinersen)
  will be evaluated with a five-point Likert Scale (from a value of 1- extremely unsatisfied to a value of 5-extremely satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico Agostino Gemelli, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Finkel RS, Mercuri E, Darras BT, Connolly AM, Kuntz NL, Kirschner J, Chiriboga CA, Saito K, Servais L, Tizzano E, Topaloglu H, Tulinius M, Montes J, Glanzman AM, Bishop K, Zhong ZJ, Gheuens S, Bennett CF, Schneider E, Farwell W, De Vivo DC; ENDEAR Study Group. Nusinersen versus Sham Control in Infantile-Onset Spinal Muscular Atrophy. N Engl J Med. 2017 Nov 2;377(18):1723-1732. doi: 10.1056/NEJMoa1702752. PMID 29091570
- [Background] Mercuri E, Darras BT, Chiriboga CA, Day JW, Campbell C, Connolly AM, Iannaccone ST, Kirschner J, Kuntz NL, Saito K, Shieh PB, Tulinius M, Mazzone ES, Montes J, Bishop KM, Yang Q, Foster R, Gheuens S, Bennett CF, Farwell W, Schneider E, De Vivo DC, Finkel RS; CHERISH Study Group. Nusinersen versus Sham Control in Later-Onset Spinal Muscular Atrophy. N Engl J Med. 2018 Feb 15;378(7):625-635. doi: 10.1056/NEJMoa1710504. PMID 29443664
- [Background] Geary RS, Yu RZ, Levin AA. Pharmacokinetics of phosphorothioate antisense oligodeoxynucleotides. Curr Opin Investig Drugs. 2001 Apr;2(4):562-73. PMID 11566019
- [Background] Zerres K, Rudnik-Schoneborn S, Forrest E, Lusakowska A, Borkowska J, Hausmanowa-Petrusewicz I. A collaborative study on the natural history of childhood and juvenile onset proximal spinal muscular atrophy (type II and III SMA): 569 patients. J Neurol Sci. 1997 Feb 27;146(1):67-72. doi: 10.1016/s0022-510x(96)00284-5. PMID 9077498
- [Background] Oskoui M, Levy G, Garland CJ, Gray JM, O'Hagen J, De Vivo DC, Kaufmann P. The changing natural history of spinal muscular atrophy type 1. Neurology. 2007 Nov 13;69(20):1931-6. doi: 10.1212/01.wnl.0000290830.40544.b9. PMID 17998484
- [Background] Kim JH, Song SY, Kim BJ. Predicting the difficulty in performing a neuraxial blockade. Korean J Anesthesiol. 2011 Nov;61(5):377-81. doi: 10.4097/kjae.2011.61.5.377. Epub 2011 Nov 23. PMID 22148085
- [Background] Fettes PD, Jansson JR, Wildsmith JA. Failed spinal anaesthesia: mechanisms, management, and prevention. Br J Anaesth. 2009 Jun;102(6):739-48. doi: 10.1093/bja/aep096. Epub 2009 May 6. PMID 19420004
- [Background] Sahin T, Balaban O, Sahin L, Solak M, Toker K. A randomized controlled trial of preinsertion ultrasound guidance for spinal anaesthesia in pregnancy: outcomes among obese and lean parturients: ultrasound for spinal anesthesia in pregnancy. J Anesth. 2014 Jun;28(3):413-9. doi: 10.1007/s00540-013-1726-1. Epub 2013 Oct 20. PMID 24141882
- [Background] Scapinelli R. Morphological and functional changes of the lumbar spinous processes in the elderly. Surg Radiol Anat. 1989;11(2):129-33. doi: 10.1007/BF02096469. PMID 2763004
- [Background] Angle P, Tang SL, Thompson D, Szalai JP. Expectant management of postdural puncture headache increases hospital length of stay and emergency room visits. Can J Anaesth. 2005 Apr;52(4):397-402. doi: 10.1007/BF03016283. PMID 15814755
- [Background] Sng BL, Lim Y, Sia AT. An observational prospective cohort study of incidence and characteristics of failed spinal anaesthesia for caesarean section. Int J Obstet Anesth. 2009 Jul;18(3):237-41. doi: 10.1016/j.ijoa.2009.01.010. Epub 2009 May 17. PMID 19450971
- [Background] Horlocker TT, McGregor DG, Matsushige DK, Schroeder DR, Besse JA. A retrospective review of 4767 consecutive spinal anesthetics: central nervous system complications. Perioperative Outcomes Group. Anesth Analg. 1997 Mar;84(3):578-84. doi: 10.1097/00000539-199703000-00021. PMID 9052305
- [Background] Vallejo MC, Phelps AL, Singh S, Orebaugh SL, Sah N. Ultrasound decreases the failed labor epidural rate in resident trainees. Int J Obstet Anesth. 2010 Oct;19(4):373-8. doi: 10.1016/j.ijoa.2010.04.002. Epub 2010 Aug 8. PMID 20696564
- [Background] Grau T, Leipold RW, Conradi R, Martin E, Motsch J. Efficacy of ultrasound imaging in obstetric epidural anesthesia. J Clin Anesth. 2002 May;14(3):169-75. doi: 10.1016/s0952-8180(01)00378-6. PMID 12031746
- [Background] Grau T, Leipold RW, Fatehi S, Martin E, Motsch J. Real-time ultrasonic observation of combined spinal-epidural anaesthesia. Eur J Anaesthesiol. 2004 Jan;21(1):25-31. doi: 10.1017/s026502150400105x. PMID 14768920
- [Background] Chin KJ, Perlas A, Chan V, Brown-Shreves D, Koshkin A, Vaishnav V. Ultrasound imaging facilitates spinal anesthesia in adults with difficult surface anatomic landmarks. Anesthesiology. 2011 Jul;115(1):94-101. doi: 10.1097/ALN.0b013e31821a8ad4. PMID 21572316
- [Background] Willschke H, Bosenberg A, Marhofer P, Willschke J, Schwindt J, Weintraud M, Kapral S, Kettner S. Epidural catheter placement in neonates: sonoanatomy and feasibility of ultrasonographic guidance in term and preterm neonates. Reg Anesth Pain Med. 2007 Jan-Feb;32(1):34-40. doi: 10.1016/j.rapm.2006.10.008. PMID 17196490
- [Background] Kallidaikurichi Srinivasan K, Iohom G, Loughnane F, Lee PJ. Conventional Landmark-Guided Midline Versus Preprocedure Ultrasound-Guided Paramedian Techniques in Spinal Anesthesia. Anesth Analg. 2015 Oct;121(4):1089-1096. doi: 10.1213/ANE.0000000000000911. PMID 26270115
- [Background] Chin KJ, Ramlogan R, Arzola C, Singh M, Chan V. The utility of ultrasound imaging in predicting ease of performance of spinal anesthesia in an orthopedic patient population. Reg Anesth Pain Med. 2013 Jan-Feb;38(1):34-8. doi: 10.1097/AAP.0b013e3182734927. PMID 23143015
- [Background] Lee PJ, Tang R, Sawka A, Krebs C, Vaghadia H. Brief report: real-time ultrasound-guided spinal anesthesia using Taylor's approach. Anesth Analg. 2011 May;112(5):1236-8. doi: 10.1213/ANE.0b013e31820ec53c. Epub 2011 Mar 3. PMID 21372276
- [Background] Karmakar MK, Li X, Ho AM, Kwok WH, Chui PT. Real-time ultrasound-guided paramedian epidural access: evaluation of a novel in-plane technique. Br J Anaesth. 2009 Jun;102(6):845-54. doi: 10.1093/bja/aep079. Epub 2009 Apr 27. PMID 19398454
- [Background] Conroy PH, Luyet C, McCartney CJ, McHardy PG. Real-time ultrasound-guided spinal anaesthesia: a prospective observational study of a new approach. Anesthesiol Res Pract. 2013;2013:525818. doi: 10.1155/2013/525818. Epub 2013 Jan 10. PMID 23365568
- [Background] Weed J, Finkel K, Beach ML, Granger CB, Gallagher JD, Sites BD. Spinal anesthesia for orthopedic surgery: a detailed video assessment of quality. Reg Anesth Pain Med. 2011 Jan-Feb;36(1):51-5. doi: 10.1097/AAP.0b013e3182030863. PMID 21455090
- [Background] Tran D, Kamani AA, Al-Attas E, Lessoway VA, Massey S, Rohling RN. Single-operator real-time ultrasound-guidance to aim and insert a lumbar epidural needle. Can J Anaesth. 2010 Apr;57(4):313-21. doi: 10.1007/s12630-009-9252-1. PMID 20196236
- [Background] Atallah MM, Demian AD, Shorrab AA. Development of a difficulty score for spinal anaesthesia. Br J Anaesth. 2004 Mar;92(3):354-60. doi: 10.1093/bja/aeh073. Epub 2004 Jan 22. PMID 14742333